CLINICAL TRIAL: NCT00361803
Title: A Phase I Study to Characterize the Pharmacokinetics of 4 mg/m2 Weekly Intravenous Topotecan in Patients With Cancer
Brief Title: Topotecan Pharmacokinetic Characterization Study
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: HYT104152
Record Dates: First submitted 2006-08-07; First posted 2006-08-09 (Estimated); Last update posted 2017-11-17 (Actual); Status verified 2017-11

CONDITIONS: Cancer
Keywords: chemotherapy; recurrent; refractory; research; cancer; pharmacokinetics
MeSH Terms: conditions — Neoplasms; Recurrence | interventions — Topotecan

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- All treated subjects (Experimental): All subjects received Topotecan, administered intravenously over 30 minutes at 4 milligrams per meter^2 weekly for 3 weeks every 28 days.
  Interventions: Drug: topotecan

INTERVENTIONS:
Drug: topotecan — topotecan

SUMMARY:
A multi-center, open label, single dose Phase I pharmacokinetic (PK) characterization of weekly IV (intravenous) topotecan given at 4mg/m2. 15 patients will be evaluated.

ELIGIBILITY:
Inclusion criteria:

* Written informed consent
* Performance status of 0, 1, or 2 on the Eastern Co-operative Oncology Group (ECOG) Scale
* Predicted life expectancy of at least 3 months
* Subjects with histologically or cytologically confirmed advanced solid tumors who have failed conventional therapy for their tumor type or have a tumor type for which no standard effective therapy exists; OR Patients for whom single-agent topotecan therapy is suitable
* At least 4 weeks since last chemotherapy, radiotherapy, biologic therapy or surgery
* Must be free of post-treatment side effects (with the exception of alopecia)
* No concurrent chemotherapy, biologic therapy or radiotherapy is allowed
* Hemoglobin = 9.0 g/dL
* WBC = 3,500/mm3 [= 3.5 x 109/L]
* Neutrophils = 1,500/mm3 [= 1.5 x 109/L]
* Platelets = 100,000/mm3 [= 100.0 x 109/L]
* Calculated creatinine clearance=60 mL/min using the Cockcroft-Gault formula
* Serum bilirubin < 2.0 mg/dL (34 µmol/L) AST, SGPT/ALT and alkaline phosphatase < 2 times the upper limit of normal if liver metastases cannot be visualized by abdominal computed tomography (CT) or magnetic resonance imaging (MRI scan)
* If liver metastases are present, subjects with < 5 times the upper limit of normal are eligible to participate

Exclusion criteria:

* Women who are pregnant or lactating
* Women subjects of childbearing potential who refuse to abstain from sexual intercourse or practice adequate contraception. Childbearing potential is defined as women who are not surgically sterilized (i.e. have not had a hysterectomy, bilateral oophorectomy [ovariectomy], or bilateral tubal ligation) or post-menopausal (i.e., documented absence of menses for one year prior to entry into the study).
* Men unwilling to abstain from sex or use effective contraception during the study and for 3 months following completion of topotecan treatment
* Subjects with uncontrolled emesis, regardless of etiology
* Active infection
* Concurrent severe medical problems unrelated to the malignancy, which would significantly limit full compliance with the study or expose the patient to extreme risk
* Treatment with another investigational drug within 30 days or five half-lives prior to entry into the study (whichever is longer)
* History of allergic reactions to compounds chemically related to topotecan.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 15 (Actual)
Dates: Start 2006-09-12 (Actual); Primary Completion 2007-08-09 (Actual); Study Completion 2007-08-09 (Actual)

PRIMARY OUTCOMES:
CL and Vss of total topotecan | Predose and at 0.25, 0.5, 0.75, 1.0, 1.5, 2.5, 4.5, 6.5, 8.5, 12, and 24 hours after the start of infusion on Day 1

SECONDARY OUTCOMES:
Cmax tmax t½ AUC(0-t) AUC(0-8) of total topotecan. Safety and tolerability will also be evaluated. | Up to 77 days

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline
Locations (1):
- GSK Investigational Site, Scottsdale, Arizona, United States

REFERENCES:
- [Background] Kurtis, KK, Jewell RC, Hartney JT, Griffin, PP, et al. Phase I study to characterize pharmacokinetics (PK) of topotecan (T) at 4 mg/m2 administered weekly as a 30-minute IV infusion. J Clin Oncol 26: 2008 (May 20 suppl; abstr 13551).
- See also: Results for study HYT104152 can be found on the GSK Clinical Study Register. — https://www.gsk-clinicalstudyregister.com/study/HYT104152?search=study&study_ids=HYT104152#rs